CLINICAL TRIAL: NCT04101201
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy of µSmin® Plus (Dietary Supplement) in Chronic Venous Insufficiency Symptoms Relief
Brief Title: Clinical Trial to Assess the Efficacy of µSmin® Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giellepi S.p.A (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CR2019/21
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Chronic Venous Disease

STUDY DESIGN:
Intervention Model Description: Diosmin is a naturally occurring flavonoid present in citrus fruits and other plants belonging to the Rutaceae family. It is used for the treatment of chronic venous insufficiency (CVI) for its pheblotonic and vaso-active properties, safety and tolerability as well.
  µSmin® Plus is a proprietary flavonoid complex with enhanced bio-efficacy. It contains highly concentrated micronized and standardized Diosmin. Highly improved bioavailability and improved oral absorption by micronization of the particles.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- µSmin® Plus (Other): µSmin® Plus is a new Micronized Diosmin Formulation for oral administration. Diosmin is extremely well tolerated and safe to use. Diosmin is safe for most people when used short-term for up to 6 months. During the 8 weeks of the clinical investigation, the subject will administer 1 tablet of µSMIN® Plus (corresponding to 450 mg of micronized diosmin) or placebo per day.
  Interventions: Dietary Supplement: µSmin® Plus
- Placebo (Placebo Comparator): It will be supplied by the Sponsor in an amount enough for the duration of the study. The subject will administer 1 tablet per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: µSmin® Plus — µSmin® Plus is a new Micronized Diosmin Formulation for oral administration. Diosmin is extremely well tolerated and safe to use. Diosmin is safe for most people when used short-term for up to 6 months. During the 8 weeks of the clinical investigation, the subject will administer 1 tablet of µSMIN® Plus (corresponding to 450 mg of micronized diosmin) or placebo per day.
  Arms: µSmin® Plus
Other: Placebo — It will be supplied by the Sponsor in an amount enough for the duration of the study. The subject will administer 1 tablet per day
  Arms: Placebo

SUMMARY:
This study evaluates treatment with the dietary supplement µSmin® Plus in a group of patients suffering from chronic venous insufficiency in comparison with a similarly-sized group of patients receiving placebo evaluated by quality of life questionnaires, VAS pain scale, CVI symptomatology, and change in the circumference of the affected leg at calf level

DETAILED DESCRIPTION:
In this study we use a dietary supplement - µSmin® Plus - for symptomatic treatment of CVI and we will monitor its impact on CVI symptoms, features, and consequences (item) of the disease listed below: limb edema, walking, daily tasks performance, pain/burning symptoms, pruritus/paresthesis, sensation of heaviness/fatigue, time wasted in the management of the disease, social burden, disease impact on self-confidence, and its impact on physical exercise/recreational activities. Results of related clinical trials were published before showing that this is an active field in clinical reasearch.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age ≥18 and ≤60 with chronic venous insufficiency;
* The chronic venous insufficiency must be graded between C2-C4 on the Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification system;
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study;
* Capable of and freely willing to provide written informed consent prior to participating in the study;
* Light smokers (<10 cigarettes per day).

Exclusion Criteria:

* Patients suffering from other or associated vascular diseases, diabetes or bleeding disorders;
* Oedema of the lower limbs of cardiac, renal or hepatic origin;
* Presence of symptoms and/or trophic disorders of arterial, metabolic, neurological or orthopedic origin including traumas, arthritis, neuropathy;
* One or more factors likely to affect venous symptoms such as recent childbirth, recent stripping, or deep or superficial venous thrombosis of the lower limbs during the previous 6 months;
* Obese subjects (BMI > 30);
* Hypersensitivity to active principles contained in the tested food supplement (diosmin);
* Patients considered smokers (≥10 cigarettes/day);
* Patients with concomitant or history of addiction to alcohol, spices or drug abuse;
* Pregnant women, nursing mothers, or women (only if childbearing potential) not using adequate methods of contraception;
* Participation in an interventional clinical study in the previous 30 days;
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed | 56 days
  Quality of life is assessed by ChronIc Venous Insuficiency quality of life Questionnaire ( CIVIQ-20 questionnaire ). The 20-item questionnaire, provides a global index and an outline of 4 quality-of-life dimensions-"pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items). Items on the CIVIQ-20 scale were scored from 1 to 5. There are 20 questions in the CIVIQ-20, each with 5 possible answers (1 to 5), the minimum possible score being 20 and the maximum 100. In order to calculate the GIS, the difference between the final score and the minimum possible score is to be divided by the difference between the theoretical maximum and minimum scores (100-20=80), multiplied by 100. A low score will correspond to greater patient comfort.
Change in the circumference of each affected leg | 56 days
  To evaluate the efficacy of the dietary supplement µSmin® Plus on ameliorating the symptoms of Chronic Venous Insufficiency in terms of change in the circumference of affected legs and quality of life, in comparison with placebo, from baseline to week 8 visit; The unit for this measurement is centimeter.

SECONDARY OUTCOMES:
Visual Analogue Scale ( VAS scale ) from 0 to 10 for pain measurements | 56 days
  Visual Analogue Scale is a straight horizontal line of 100 mm. The ends are defined as the extreme limits of the pain (symptom, pain, health) orientated from the left (worst) to the right (best). Using a ruler, the score is determined by measuring the distance in millimeters on the 10 centimeters line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity and a low score indicates a low pain intensity.
Symptoms relief assessed by Venous Clinical Severity Score (VCSS) questionnaire | 56 days
  Venous Clinical Severity Score use the progressive ranking of severity, while weighting the upper levels representing the more severe presentations of Chronical Venous Disease. The lowest possible score is 0=absent meaning that the patient has no symptoms and the highest possible score is 30=sever meaning that the patient has a very severe venous symptoms.
Investigator Global Assessment of the efficacy by scoresproduct | 56 days
  Efficacy of treatment: Percentage of physicians who rated 1= excellent, 2 = good, 3= fair, 4= poor
Patient Global Assessment of the efficacy by scores | 56 days
  Patients satisfaction: 1= very satisfied, 2= satisfied, 3 = adequate, 4= unsatisfied, 5 = very unsatisfied
Percentage of subjects who would want to continue with µSmin® Plus. | 56 days
  By this outcome we want to find out the percentage of patients who will want to continue with µSmin® Plus.
Percentage of subjects who experienced symptoms relief | 56 days
  Percentage of subjects who experienced symptoms relief within the first week of intake, within 2 weeks of intake, or more than 2 weeks of intake;
Treatment compliance | 56 days
  Variable medication possession ratio (VMPR) will be used to calculate the compliance (or adherence) to the treatment in the two groups collected by diary card and used and unused products
AE/SAE incidence | 56 days
  Evaluation of safety during all the study period through AE/SAE collection
Investigator Global Assessment of Safety (IGAS): | 56 days
  Investigator Global Assessment of Safety (IGAS): using the 4-point scale:1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated at the last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Doina Rosu, MD, Principal Investigator — SCM Dr. Rosu
Locations (1):
- SCM Gados, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Robertson L, Evans C, Fowkes FG. Epidemiology of chronic venous disease. Phlebology. 2008;23(3):103-11. doi: 10.1258/phleb.2007.007061. PMID 18467617
- [Background] Onida S, Davies AH. Predicted burden of venous disease. Phlebology. 2016 Mar;31(1 Suppl):74-9. doi: 10.1177/0268355516628359. PMID 26916773
- [Background] Carpentier PH, Maricq HR, Biro C, Poncot-Makinen CO, Franco A. Prevalence, risk factors, and clinical patterns of chronic venous disorders of lower limbs: a population-based study in France. J Vasc Surg. 2004 Oct;40(4):650-9. doi: 10.1016/j.jvs.2004.07.025. PMID 15472591
- [Background] Malone PC, Agutter PS. To what extent might deep venous thrombosis and chronic venous insufficiency share a common etiology? Int Angiol. 2009 Aug;28(4):254-68. PMID 19648868
- [Background] Russo R, Mancinelli A, Ciccone M, Terruzzi F, Pisano C, Severino L. Pharmacokinetic Profile of microSMIN Plus, a new Micronized Diosmin Formulation, after Oral Administration in Rats. Nat Prod Commun. 2015 Sep;10(9):1569-72. PMID 26594761
- [Background] Russo R, Chandradhara D, De Tommasi N. Comparative Bioavailability of Two Diosmin Formulations after Oral Administration to Healthy Volunteers. Molecules. 2018 Aug 29;23(9):2174. doi: 10.3390/molecules23092174. PMID 30158431
- [Background] Belczak SQ, Sincos IR, Campos W, Beserra J, Nering G, Aun R. Veno-active drugs for chronic venous disease: A randomized, double-blind, placebo-controlled parallel-design trial. Phlebology. 2014 Aug;29(7):454-60. doi: 10.1177/0268355513489550. Epub 2013 May 16. PMID 23761871
- [Background] Zolotukhin IA, Seliverstov EI, Shevtsov YN, Avakiants IP, Nikishkov AS, Tatarintsev AM, Kirienko AI. Prevalence and Risk Factors for Chronic Venous Disease in the General Russian Population. Eur J Vasc Endovasc Surg. 2017 Dec;54(6):752-758. doi: 10.1016/j.ejvs.2017.08.033. Epub 2017 Oct 12. PMID 29031868
- [Background] Vuylsteke ME, Thomis S, Guillaume G, Modliszewski ML, Weides N, Staelens I. Epidemiological study on chronic venous disease in Belgium and Luxembourg: prevalence, risk factors, and symptomatology. Eur J Vasc Endovasc Surg. 2015 Apr;49(4):432-9. doi: 10.1016/j.ejvs.2014.12.031. Epub 2015 Feb 18. PMID 25701071
- [Background] Lichota A, Gwozdzinski L, Gwozdzinski K. Therapeutic potential of natural compounds in inflammation and chronic venous insufficiency. Eur J Med Chem. 2019 Aug 15;176:68-91. doi: 10.1016/j.ejmech.2019.04.075. Epub 2019 May 6. PMID 31096120
- [Background] Rabe E, Guex JJ, Morrison N, Ramelet AA, Schuller-Petrovic S, Scuderi A, Staelens I, Pannier F. Treatment of chronic venous disease with flavonoids: recommendations for treatment and further studies. Phlebology. 2013 Sep;28(6):308-19. doi: 10.1177/0268355512471929. Epub 2013 May 6. PMID 23395842
- [Background] Lebeau J, Furman C, Bernier JL, Duriez P, Teissier E, Cotelle N. Antioxidant properties of di-tert-butylhydroxylated flavonoids. Free Radic Biol Med. 2000 Nov 1;29(9):900-12. doi: 10.1016/s0891-5849(00)00390-7. PMID 11063915
- [Background] Panche AN, Diwan AD, Chandra SR. Flavonoids: an overview. J Nutr Sci. 2016 Dec 29;5:e47. doi: 10.1017/jns.2016.41. eCollection 2016. PMID 28620474
- [Background] Bakhtiari M, Panahi Y, Ameli J, Darvishi B. Protective effects of flavonoids against Alzheimer's disease-related neural dysfunctions. Biomed Pharmacother. 2017 Sep;93:218-229. doi: 10.1016/j.biopha.2017.06.010. Epub 2017 Jun 20. PMID 28641164
- [Background] Milano G, Leone S, Fucile C, Zuccoli ML, Stimamiglio A, Martelli A, Mattioli F. Uncommon serum creatine phosphokinase and lactic dehydrogenase increase during diosmin therapy: two case reports. J Med Case Rep. 2014 Jun 16;8:194. doi: 10.1186/1752-1947-8-194. PMID 24934505
- [Background] Heinen M, Borm G, van der Vleuten C, Evers A, Oostendorp R, van Achterberg T. The Lively Legs self-management programme increased physical activity and reduced wound days in leg ulcer patients: Results from a randomized controlled trial. Int J Nurs Stud. 2012 Feb;49(2):151-61. doi: 10.1016/j.ijnurstu.2011.09.005. Epub 2011 Sep 28. PMID 21959100
- [Background] Martinez-Zapata MJ, Vernooij RW, Uriona Tuma SM, Stein AT, Moreno RM, Vargas E, Capella D, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2016 Apr 6;4(4):CD003229. doi: 10.1002/14651858.CD003229.pub3. PMID 27048768
- [Background] Kakkos SK, Nicolaides AN. Efficacy of micronized purified flavonoid fraction (Daflon(R)) on improving individual symptoms, signs and quality of life in patients with chronic venous disease: a systematic review and meta-analysis of randomized double-blind placebo-controlled trials. Int Angiol. 2018 Apr;37(2):143-154. doi: 10.23736/S0392-9590.18.03975-5. Epub 2018 Jan 31. PMID 29385792
- [Background] Wilson D, Wakefield M, Owen N, Roberts L. Characteristics of heavy smokers. Prev Med. 1992 May;21(3):311-9. doi: 10.1016/0091-7435(92)90030-l. PMID 1614993
- [Background] Freag MS, Elnaggar YS, Abdallah OY. Lyophilized phytosomal nanocarriers as platforms for enhanced diosmin delivery: optimization and ex vivo permeation. Int J Nanomedicine. 2013;8:2385-97. doi: 10.2147/IJN.S45231. Epub 2013 Jul 3. PMID 23861584